CLINICAL TRIAL: NCT01089140
Title: Blood Loss and Transfusion Requirement in Pediatric Patients With Non-Idiopathic Scoliosis Treated With Tranexamic Acid Undergoing Posterior Spinal Instrumentation and Fusion.
Brief Title: Non-Idiopathic Scoliosis Treated With Tranexamic Acid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate number of potential participants
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Tara Der, Staff Anaesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1000013524
Record Dates: First submitted 2010-03-11; First posted 2010-03-18 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Non-idiopathic Scoliosis
Keywords: pediatrics; scoliosis; tranexamic acid; Investigating non-idiopathic scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- . Tranexamic acid low dose 10 mg/kg (Experimental)
  Interventions: Drug: Tranexamic acid 10mg/kg/hr
- Tranexamic acid 100mg/kg (Experimental)
  Interventions: Drug: Tranexamic acid 100 mg/kg/h infusion
- Saline Placebo (Placebo Comparator)
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Tranexamic acid 10mg/kg/hr — Tranexamic acid is a synthetic antifibrinolytic drug that competitively inhibits the lysine binding sites of plasminogen, plasmin, and tissue plasminogen activator
  Other Names: TXA
  Arms: . Tranexamic acid low dose 10 mg/kg
Drug: Tranexamic acid 100 mg/kg/h infusion — Tranexamic acid is a synthetic antifibrinolytic drug that competitively inhibits the lysine binding sites of plasminogen, plasmin, and tissue plasminogen activator.
  Other Names: TXA
  Arms: Tranexamic acid 100mg/kg
Drug: Saline solution — Saline placebo
  Arms: Saline Placebo

SUMMARY:
Investigation of tranexamic acid (TXA) for reducing perioperative blood loss and transfusion requirement in pediatric patients with secondary scoliosis undergoing posterior spinal fusion.

DETAILED DESCRIPTION:
To investigate whether tranexamic acid (TXA) reduces perioperative blood loss and transfusion requirement in pediatric patients with secondary scoliosis undergoing posterior spinal fusion.In addition determination of the optimal TXA dosing for perioperative reduction of blood loss and transfusion requirement as well as to evaluate use of thromboelastography (TEG) as a measure of coagulation and fibrinolysis in pediatric patients with secondary scoliosis undergoing posterior spinal fusion (this may help guide blood product therapy).

The investigation will determine the effects of TXA on the TEG profile and whether plasminogen activator inhibitor-1 (PAI-1) level affects bleeding and transfusion requirement during scoliosis surgery. Finally to investigate whether PAI-1 level affects bleeding in response to TXA during scoliosis surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Children with secondary scoliosis undergoing posterior spinal fusion

Exclusion Criteria:

1. Known bleeding disorder as this may increase the risk of bleeding
2. Current antifibrinolytic therapy as these patients may bleed less
3. Patient or family history of thromboembolic disease as there may be potential risk of thrombosis
4. Use of NSAIDS within 5 days of surgery as this may increase the risk of bleeding
5. Known allergy to TXA
6. History of renal insufficiency as TXA is renally excreted
7. Colour vision disturbance

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss and transfusion requirement | 8 hours

SECONDARY OUTCOMES:
Thromboelastography (TEG): TEG monitors coagulation of blood samples in vitro to produce a complete picture of clot formation, strength and dissolution (i.e. fibrinolysis). | After Induction- Prior to Drug Administration, Immediately after Bolus Dose
Plasminogen Activator Inhibitor-1 | Baseline -Immediately after induction and prior to administration of study drug
  Different genotypes for the plasminogen activator inhibitor-1 (PAI-1) gene may have varying degrees of bleeding. PAI-1 inhibits the transformation of plasminogen to plasmin thereby decreasing plasmin-induced fibrinolysis. Thus, PAI-1 promotes clot stability.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Der, M.sc. MD.,(FRCPC), Principal Investigator — Hospital for SickkIds
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada